CLINICAL TRIAL: NCT00189215
Title: Long-Term Cognitive Decline After Coronary Artery Bypass Grafting: is Off-Pump Surgery Beneficial?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: International Anesthesia Research Society (IARS) (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: WOM protocol 98/009-O
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2007-12-04 (Estimated); Status verified 2005-03

CONDITIONS: Coronary Artery Disease; Cardiopulmonary Bypass; Cognition Disorders
Keywords: coronary artery disease; cardiopulmonary bypass; cognition disorders
MeSH Terms: conditions — Coronary Artery Disease; Cognition Disorders

INTERVENTIONS:
Device: cardiac stabilizer instead of cardiopulmonary bypass

SUMMARY:
Coronary artery bypass surgery is associated with postoperative cognitive decline, which has largely been attributed to the use of the heart lung machine. We hypothesized that long-term cognitive outcome may improve by avoiding the heart lung machine. The objective of the present study is to compare the effect of coronary bypass surgery with and without heart lung machine on cognitive and clinical outcome, five years after surgery.

DETAILED DESCRIPTION:
Background:

Coronary artery bypass surgery is associated with postoperative cognitive decline, which has largely been attributed to the use of cardiopulmonary bypass (CPB). A large recent study by Newman et al demonstrated that the incidence of cognitive decline was 24% at six months after surgery, but it increased to 42% at five years. In the recently conducted Octopus Randomized Trial, cognitive decline at three months after surgery was present in 29% of the patients operated with CPB. In the patients operated without CPB, the incidence was 21%, i.e. only slightly better.

Hypothesis:

Improvement of cognitive outcome by avoiding cardiopulmonary bypass will become more apparent five years after surgery, compared to three months after surgery.

Study objectives:

The objective of the present study is to compare the effect of coronary bypass surgery with and without cardiopulmonary bypass on cognitive and clinical outcome, five years after surgery.

Methods:

The 281 participants of the Octopus Study, who were operated on between March 1998 and August 2000 and randomized to off-pump or on-pump coronary bypass surgery, will be invited for an additional assessment of their cognitive and clinical status and quality of life, five years after surgery. Patients will undergo a battery of ten neuropsychologic tests to determine their cognitive status. Clinical status will be assessed by an interview. Questionnaires will be used to measure quality of life.

ELIGIBILITY:
Inclusion Criteria:

* indication for (first-time) coronary artery bypass surgery
* off-pump CABG considered technically possible

Exclusion Criteria:

* concomitant valve surgery
* unable to complete neuropsychological testing
* life expectancy less than 1 year

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 280
Dates: Start 1998-03; Study Completion 2005-12

PRIMARY OUTCOMES:
cognitive decline 5 year after the index treatment

SECONDARY OUTCOMES:
-freedom from cardiovascular events (i.e. mortality, stroke, myocardial infarction, re-CABG, or PTCA
-recurrence of angina
-use of anti-anginal drugs
-quality of life (SF-36 and EuroQuol

CONTACTS AND LOCATIONS:
Overall Officials: Cor J Kalkman, MD, PhD, Study Director — UMC Utrecht, The Netherlands
Locations (1):
- University Medical Center, Department of Anesthesiology, Utrecht, Utrecht, Netherlands

REFERENCES:
- [Background] van Dijk D, Nierich AP, Eefting FD, Buskens E, Nathoe HM, Jansen EW, Borst C, Knape JT, Bredee JJ, Robles de Medina EO, Grobbee DE, Diephuis JC, de Jaegere PP. The Octopus Study: rationale and design of two randomized trials on medical effectiveness, safety, and cost-effectiveness of bypass surgery on the beating heart. Control Clin Trials. 2000 Dec;21(6):595-609. doi: 10.1016/s0197-2456(00)00103-3. PMID 11146152
- [Result] Van Dijk D, Jansen EW, Hijman R, Nierich AP, Diephuis JC, Moons KG, Lahpor JR, Borst C, Keizer AM, Nathoe HM, Grobbee DE, De Jaegere PP, Kalkman CJ; Octopus Study Group. Cognitive outcome after off-pump and on-pump coronary artery bypass graft surgery: a randomized trial. JAMA. 2002 Mar 20;287(11):1405-12. doi: 10.1001/jama.287.11.1405. PMID 11903027
- [Result] Nathoe HM, van Dijk D, Jansen EW, Suyker WJ, Diephuis JC, van Boven WJ, de la Riviere AB, Borst C, Kalkman CJ, Grobbee DE, Buskens E, de Jaegere PP; Octopus Study Group. A comparison of on-pump and off-pump coronary bypass surgery in low-risk patients. N Engl J Med. 2003 Jan 30;348(5):394-402. doi: 10.1056/NEJMoa021775. PMID 12556542